CLINICAL TRIAL: NCT04033484
Title: Pelvic Floor Reconstruction Using Biological Mesh With Negative Pressure Wound Therapy Following Extralevator Abdominoperineal Excision
Brief Title: Pelvic Floor Reconstruction Using Biological Mesh With Negative Pressure Wound Therapy Following ELAPE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zhen Jun Wang, Chairman of General Surgery, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bio-NEST 01
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Perineal Wound Complications After ELAPE
Keywords: extralevator abdominoperineal excision; Perineal wound healing; negative pressure wound therapy; biological mesh
MeSH Terms: interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biological Mesh (Active Comparator): Using biological mesh to recnostruct the pelvic floor following ELAPE
  Interventions: Procedure: Negative Pressure Wound Therapy
- Biological Mesh With Negative Pressure Wound Therapy (Experimental): Using biological mesh compined with negative pressure wound therapy to recnostruct the pelvic floor following ELAPE
  Interventions: Procedure: Negative Pressure Wound Therapy

INTERVENTIONS:
Procedure: Negative Pressure Wound Therapy — The perineal wound was reconstructed with biologic mesh after ELAPE. The subcutaneous adipose layer was closed with 2/0 vicryl sutures, and a suction drain was left in the deep layer. The subcuticular layer and skin were closed with 3/0 vicryl mattress sutures and the negative pressure system applied at 80 mmHg

SUMMARY:
Perineal wound healing is a significant challenge after extralevator abdominoperineal excision (ELAPE) due to a high rate of wound breakdown. And it was proved that neoadjuvant radiotherapy significantly increases perineal wound problems after abdominoperineal resection for rectal cancer. Negative pressure therapy has proven benefits in open wounds, and recently a negative pressure system has been developed for use on closed wounds at high risk of breakdown. A systematic review suggested a significant decrease in perineal wound complications when using incisional negative pressure wound therapy was demonstrated, with surgical site infection rates as low as 9% (vs 41% in control groups). The review suggested that incisional negative pressure wound therapy decreases perineal wound complications after abdominoperineal resection. Prospective study also suggested that after ELAPE the application of a negative pressure system to the perineal wound closed with biologic mesh may reduce perineal wound complications. The aim of the present study was to determine whether negative pressure therapy combined with biological mesh compared with biological mesh alone after ELAPE could improve wound healing.

ELIGIBILITY:
Inclusion Criteria:

1. Rectal cancer within 4 cm of the anal verge
2. T3 or T4, as determined by pre-operative MRI examination; patient did receive neoadjuvant chemoradiotherapy
3. Absence of distant metastases
4. Absence of intestinal obstruction

Exclusion Criteria:

1. T1-T2, as determined by pre-operative MRI before neoadjuvant chemoradiotherapy
2. Distant metastases
3. Intestinal obstruction
4. Pregnancy or lactating
5. Contraindications to surgery
6. A mental disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
perineal wound complications | 6 months after operation
  perineal wound complications after pelvic floor reconstruction following ELAPE

CONTACTS AND LOCATIONS:
Locations (1):
- Zhen Jun. Wang, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Perineal wound healing is a significant challenge after extralevator abdominoperineal excision (ELAPE) due to a high rate of wound breakdown. And it was proved that neoadjuvant radiotherapy significantly increases perineal wound problems after abdominoperineal resection for rectal cancer. Negative pressure therapy has proven benefits in open wounds, and recently a negative pressure system has been developed for use on closed wounds at high risk of breakdown. Prospective study also suggested that after ELAPE the application of a negative pressure system to the perineal wound closed with biologic mesh may reduce perineal wound complications. The aim of the present study was to determine whether negative pressure therapy combined with biological mesh compared with biological mesh alone after ELAPE could improve wound healing.
Supporting Information: Study Protocol
Time Frame: 2019.07.1-2021.07.31
Access Criteria: Inclusion criteria
  1. Tumor within 4 cm of the anal verge
  2. T3 or T4, as determined by pre-operative MRI examination; patient did receive neoadjuvant chemoradiotherapy
  3. Absence of distant metastases
  4. Absence of intestinal obstruction